CLINICAL TRIAL: NCT06689436
Title: A Pivotal, Randomized, Single-dose, Open-label, Four-Way Crossover, BE Study of TAH3311 (Apixaban ODF) Under Fasted and Fed Conditions vs. ELIQUIS® Oral Tablet Under Fasted Condition in Healthy Volunteers
Brief Title: Pivotal BE Study of TAH3311 ODF vs ELIQUIS® Tablet Under Fasted Condition in Healthy Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TAHO Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: TAH3311-CP-2301
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Random Allocation; Intermittent Fasting; Enteral Feeding
Keywords: Crossover Design; Therapeutic Equivalency
MeSH Terms: conditions — Intermittent Fasting | interventions — apixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- 5 mg Apixaban Oral Dissolving Film (fasting) (Experimental): Treatment T1: Subject will receive a single dose of 5 mg Apixaban Oral Dissolving Film under fasting condition
  Interventions: Drug: 5 mg Apixaban Oral Dissolving Film (fasting)
- 5 mg Apixaban Oral Dissolving Film (fed) (Experimental): Treatment T2: Subject will receive a single dose of 5 mg Apixaban Oral Dissolving Film under fed condition.
  Interventions: Drug: 5 mg Apixaban Oral Dissolving Film (fed)
- 5 mg Apixaban Oral Tablet (US RS/RLD) (Active Comparator): Treatment R1: Subject will receive a single dose of 5 mg Apixaban Oral Tablet (US RS/RLD) under fasting condition.
  Interventions: Drug: 5 mg Apixaban Oral Tablet (US RS/RLD)
- 5 mg Apixaban Oral Tablet (EU product) (Active Comparator): Treatment R2: Subject will receive a single dose of 5 mg Apixaban Oral Tablet (EU product)) under fasting condition.
  Interventions: Drug: 5 mg Apixaban Oral Tablet (EU product)

INTERVENTIONS:
Drug: 5 mg Apixaban Oral Dissolving Film (fasting) — Single dose of 5 mg Apixaban Oral Dissolving Film will be administered orally after at least 10 hours overnight fast
  Other Names: TAH3311 ODF
  Arms: 5 mg Apixaban Oral Dissolving Film (fasting)
Drug: 5 mg Apixaban Oral Dissolving Film (fed) — Single dose of 5 mg Apixaban Oral Dissolving Film will be administered orally at 30 minutes after the start of a standardized high-fat, high-calorie breakfast that is preceded by at least 10 hours overnight fast
  Arms: 5 mg Apixaban Oral Dissolving Film (fed)
Drug: 5 mg Apixaban Oral Tablet (US RS/RLD) — Single dose of 5 mg Apixaban Oral Tablet (US RS/RLD) will be administered orally after at least 10 hours overnight fast
  Other Names: ELIQUIS® (US RS/RLD)
  Arms: 5 mg Apixaban Oral Tablet (US RS/RLD)
Drug: 5 mg Apixaban Oral Tablet (EU product) — Single dose of 5 mg Apixaban Oral Tablet (EU product) will be administered orally after at least 10 hours overnight fast
  Arms: 5 mg Apixaban Oral Tablet (EU product)

SUMMARY:
This single-dose, open-label, randomized, four-way crossover study evaluates the pharmacokinetics, safety, and tolerability of TAH3311 5 mg in healthy volunteers under fasted and fed conditions.

DETAILED DESCRIPTION:
Eligible subjects will be enrolled in the study across four sequences (anticipate 15 subjects per sequence). This study will have three phases: Screening Phase, Treatment Phase, and Follow-Up Phase. Subjects will be randomized 1:1:1:1 to receive TAH3311 ODF 5 mg under fasted (T1) and fed conditions (T2) and ELIQUIS® 5 mg (US RS/RLD [R1] and EU product [R2]) under fasted condition via one of the four sequences with serial PK sampling from 90 minutes pre-dose to 48 hours post-dose. The duration of each treatment period is 4 days, with a 7±2 days washout in between of the treatment administration. The follow-up period will be 7±3 days after the last treatment dosing.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL the following criteria at time of Screening:

1. Subject is a male or female, 18-80 years of age, inclusive.
2. Weight within the BMI of 18-32 kg/m2 inclusive and weighs at least 60 kg.
3. Subject is willing and able to participate in all scheduled visits including follow up, treatment plan, laboratory tests and other study procedures according to clinical protocol.
4. The subject is in good health and has no medical condition of clinical significance or that may impact the outcome of the study, as determined by the investigator.
5. The subject is able to understand the nature of the study and any potential hazards associated with participating in it.
6. Subject doesn't have any relevant dietary restrictions, as determined by the Investigator, and is willing to consume a high-fat, high-calorie breakfast and other standard meals provided during the treatment periods of the study, and to comply with the fasting conditions required by the study design.
7. The subject is able to communicate satisfactorily with the investigator and to participate in, and comply with, the requirements of the study.
8. The subject is willing to provide written informed consent to participate in the study after reading the informed consent form and the information provided and has had the opportunity to discuss the study with the investigator or designee.
9. If female and not infertile (defined below), the subject must agree for the duration of the study to use one of the following forms of contraception 1) systemic hormonal treatment 2) an intrauterine device (IUD) which was implanted at least 2 months prior to screening or 3) "double-barrier" contraception (condom, diaphragm and spermicide are each considered a barrier). Females are considered to be infertile if they are either a) surgically sterile or b) have had spontaneous amenorrhea for at least the last 2 years and at least 2 years after the onset of amenorrhea while not receiving hormone replacement therapy and had a Follicle-Stimulating Hormone (FSH) level greater than 40 mIU/mL and an estradiol level less than 30 pg/mL.
10. Male subjects who are not surgically sterile must agree to use appropriate contraceptive measures and agree to not impregnate a female partner(s) and not to donate sperm throughout the entire study, including the washout periods, and for 30 days after the last study drug administration. Examples of acceptable methods of contraception include a double-barrier method of contraception (e.g., condom with spermicide). Other forms of contraception may be acceptable, at the discretion of the Investigator.

Exclusion Criteria:

Subjects meeting ANY of the following criteria at time of Screening will be excluded from enrollment:

1. The subject has a history of severe allergic or anaphylactic reactions.
2. The subject has a known allergy or hypersensitivity to Apixaban, or history of any food or drug hypersensitivity or intolerance which in the opinion of the Investigator, would compromise the safety of the subject or the study.
3. Current tongue piercing or other piercings in the mouth, including lips and cheeks which have studs/rings, etc. or where the piercing wound is not completely closed or any tongue or other oral deformities that may affect the absorption of the drug product.
4. The subject has a medical history or current evidence of system disorders, organ dysfunction especially cardiovascular disorders (e.g., atrial fibrillation), renal or hepatic disorders which in the opinion of the Investigator, would compromise the safety of the subject or the study.
5. Female subjects who are pregnant or lactating.
6. The subject has a Family history of sudden cardiac death.
7. The subject has a history of blood clots or bleeding disorders (e.g., bleeding diathesis [tendency to bleed or bruise easily]), stroke, or active pathological bleeding.
8. The subject has a clinically significant history or are currently at risk for arterial or venous thromboembolic events (e.g., transient ischemic attack, cerebrovascular accident, myocardial infarction, retinal artery occlusion or retinal vein thrombosis, pulmonary embolism, deep vein thrombosis, antiphospholipid syndrome), as determined by the Investigator.
9. The subject has had an acute infection within 2 weeks before screening or at any time between screening and check-in including, but not limited to, history, signs, or symptoms of a common cold (e.g., mild rhinorrhea), untreated oral/dental abnormalities (e.g., untreated dental caries as determined by examination of the mouth), or untreated disruption of the skin.
10. The subject has a positive test for human immunodeficiency virus (HIV) types 1 or 2, Hepatitis B surface antigen or Hepatitis C antibody (HCV) at screening.
11. Subject has any active infection requiring systemic therapy at the time of screening, which is considered clinically significant per the Principial Investigator.
12. The investigator determined the subject has a history of or ongoing chronic or recurrent infectious disease (e.g., infected indwelling prosthesis, osteomyelitis, chronic sinusitis)
13. Drug or alcohol addiction requiring treatment in the 12 months before initial dosing.
14. History of excessive alcohol consumption (on average more than 14 units of alcohol/week; 1 unit = 12 oz. beer, 6 oz. wine, 1 shot [1.5 oz.] of liquor) during the past 12 months.
15. The subject has taken any medications (including herbal remedies) known to significantly induce or inhibit drug metabolizing enzymes (especially inhibitors and inducers of CYP3A4 and P-gp such as ketoconazole, itraconazole, ritonavir, clarithromycin, rifampin, phenytoin, carbamazepine, St. John's Wort, etc.) within 30 days before initial dosing and other medications deemed acceptable by the Principal Investigator.
16. Clinically significant history or presence of gastrointestinal disease (e.g., bleeding, perforation, or fistulas) or malabsorption, as determined by the Investigator.
17. The subject has participated in another clinical study of a new investigational drug or has received an investigational drug within 28 days or 5 half-lives (if available) before study drug administration, whichever is longer.
18. Anticipating undergoing surgery or medical/dental procedure, receiving neuraxial anesthesia (spinal/epidural anesthesia), or undergoing spinal puncture during the study or within 7 days after study completion.
19. Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days before initial dosing.
20. Subject has difficulty swallowing, as determined by the investigator.
21. Subject has a prosthetic heart valve.
22. Subject has abnormal prothrombin time (PT) and activated partial thromboplastin time (aPTT).
23. The subject has serum creatinine ≥1.5 mg/dL
24. eGFR<90 mL/min/1.73 m2; obtained from the clinical laboratory tests performed at screening.
25. Use of drugs affecting hemostasis such as aspirin and other antiplatelet agents, other anticoagulants, heparin, thrombolytic agents, selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), and nonsteroidal anti-inflammatory drugs (NSAIDs) within 14 days before initial dosing.
26. Positive test results for drugs of abuse or cotinine at screening
27. The subject is unable to participate in, or successfully complete, the study, in the opinion of the investigator, because the subject is any of the following:

    * Mentally or legally incapacitated, or unable to give consent for any reason
    * Unlikely to cooperate or comply with the clinical study protocol or is unsuitable for any other reason

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-11-16 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of Apixaban for TAH3311 Oral Dissolving Film (ODF) under fasted and fed conditions | From enrollment to the end of treatment at 10 weeks
Peak Plasma Concentration (Cmax) of Apixaban for ELIQUIS® 5 mg Oral Tablet under fasted condition | From enrollment to the end of treatment at 10 weeks
Area under the plasma concentration curve from time zero to last sampling time (AUC0-t) of Apixaban for TAH3311 Oral Dissolving Film (ODF) under fasted and fed conditions | From enrollment to the end of treatment at 10 weeks
Area under the plasma concentration curve from time zero to last sampling time (AUC0-t) of Apixaban for ELIQUIS® 5 mg Oral Tablet under fasted condition | From enrollment to the end of treatment at 10 weeks
Area under the plasma concentration curve from time zero to infinity (AUC0-∞) of Apixaban for TAH3311 Oral Dissolving Film (ODF) under fasted and fed conditions | From enrollment to the end of treatment at 10 weeks
Area under the plasma concentration curve from time zero to infinity (AUC0-∞) of Apixaban for ELIQUIS® 5 mg Oral Tablet under fasted condition | From enrollment to the end of treatment at 10 weeks

SECONDARY OUTCOMES:
Area under the plasma concentration curve from time zero to infinity (AUC0-∞) of Apixaban for TAH3311 Oral Dissolving Film (ODF) under fasted and fed conditions | From enrollment to the end of treatment at 10 weeks
Area under the plasma concentration curve from time zero to infinity (AUC0-∞) of Apixaban for ELIQUIS® 5mg Oral Tablets (for the EU product) under fasted conditions | From enrollment to the end of treatment at 10 weeks
Obtaining specific pharmacokinetic parameters for Apixaban following single dose administration under fasted and fed conditions: | From enrollment to the end of treatment at 10 weeks
  The specific PK parameters to be calculated include at least:
  * Apparent terminal elimination half-life (t1/2)
  * Time to maximum observed plasma drug concentration (Tmax)

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany A Bradley, MD, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, USA, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided